CLINICAL TRIAL: NCT07139522
Title: The Efficacy of Dexamethasone Versus Magnesium Sulphate as an Adjuvant to Bupivacaine in Ultrasound Guided Erector Spinae Plane Block for Postoperative Analgesia in Elective Caesarean Section Under Spinal Anesthesia: A Randomized Controlled Trial.
Brief Title: Dexamethasone Versus Magnesium Sulphate as an Adjuvant to Bupivacaine in Ultrasound Guided Erector Spinae Plane Block for Postoperative Analgesia in Elective Caesarean Section Under Spinal Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Esmaeel Sayed Farrag, Assistant Lecturer of Anesthesia, Surgical ICU and Pain Medicine, Faculty of Medicine, Cairo University, Cairo, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-344-2023
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Dexamethasone; Magnesium Sulphate; Adjuvant; Ultrasound; Erector Spinae Plane Block; Postoperative Analgesia; Cesarean Section; Spinal Anesthesia
MeSH Terms: interventions — Bupivacaine; Dexamethasone; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Patients will receive 20 ml 0.25% isobaric bupivacaine.
  Interventions: Drug: Bupivacaine
- Dexamethasone group (Experimental): Patients will receive 20 ml of (0.25% isobaric bupivacaine and 4mg of dexamethasone).
  Interventions: Drug: Dexamethasone
- Magnesium group (Experimental): Patients will receive 20 ml of (0.25% isobaric bupivacaine and 200mg of magnesium sulphate).
  Interventions: Drug: Magnesium sulphate

INTERVENTIONS:
Drug: Bupivacaine — Patients will receive 20 ml of 0.25% isobaric bupivacaine.
  Arms: Control group
Drug: Dexamethasone — Patients will receive 20 ml of (0.25% isobaric bupivacaine and 4mg of dexamethasone).
  Arms: Dexamethasone group
Drug: Magnesium sulphate — Patients will receive 20 ml of (0.25% isobaric bupivacaine and 200mg of magnesium sulphate).
  Arms: Magnesium group

SUMMARY:
This study aims to compare the efficacy of adding dexamethasone and magnesium sulfate as an adjuvant to bupivacaine in bilateral erector spinae block in postoperative pain control in patients undergoing caesarean section under spinal anesthesia.

DETAILED DESCRIPTION:
Caesarean section (CS) is the most common abdominal surgery among women worldwide. Inadequately treated postoperative pain can contribute significantly to morbidity of surgical patients, resulting in the delay of patients' recovery and ability to return to daily functional activities, increased incidence of chronic pain, and post-traumatic stress syndrome.

The ultrasound-guided erector spinae plane (ESP) block is a recently described interfascial paraspinal plane technique that was initially used by Forero et al. for providing thoracic analgesia when performed at the level of T5 transverse process. Since the pain experienced after caesarean delivery using a Pfannenstiel incision has both a somatic and visceral component.

Magnesium sulfate (MgSO4) may be helpful as an analgesic adjuvant in regional anesthesia because it improves and prolongs the analgesic effect of local anesthetics.

Dexamethasone is a potent glucocorticoid medication commonly used as an adjuvant to reduce postoperative pain. The mechanisms of perineurally administered dexamethasone are likely attributed to complex interactions, including direct inhibition of signal transmission in nociceptive C fibres, local vasoconstriction, and reduced local inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 35 years.
* Full-term, singleton, pregnant women.
* American Society of Anesthesiologists (ASA) physical status II.
* Scheduled for elective cesarean delivery under spinal anesthesia.

Exclusion Criteria:

* Refusal of the patient.
* Emergency caesarean sections.
* Patients having chronic diseases as asthma, cardiovascular disorders (Significant arrhythmias, Severe Valvular diseases, congenital heart diseases, ischemic heart disease, cardiomyopathy, deep venous thrombosis ,and pulmonary embolism)
* Renal impairment (Creatinine level ≥ 2mg/dl, urea ≥ 25mg/dL), liver impairment [Alanine aminotransferase (ALT) < 45 U/L, Aspartate aminotransferase (AST) < 45 U/L].
* Allergy to the drug enrolled in the study.
* Body mass index (BMI) ≥ 35 kg/m2.
* Hypertensive disorders of pregnancy.
* Contraindication to spinal anesthesia, such as coagulopathy [platelet count <150.000, international normalized ratio (INR) > 1.2], or local infection.
* Requirement for conversion to general anesthesia after spinal anesthesia will also be excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women undergoing elective cesarean section
Enrollment: 150 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to first analgesic requirement | 24 hours postoperatively
  Time to first analgesic requirement in the following 24 hours after cesarean delivery. It is the time elapsed between performing the assigned intervention and first morphine requirement.

SECONDARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be recorded at 1, 2, 4, 6,18 and 24 h postoperatively.
Obstetric Quality of Recovery | 24 hours postoperatively
  Obstetric Quality of Recovery (ObsQore) aims to measure functional recovery at 24 hours postpartum quantitatively. It includes 11 questions on a 0 to 11 scale, and the results are tabulated out of 100. The higher the overall score out of 100, the better quality of recovery a patient is experiencing, aimed at pain management, the adverse effects of narcotics, and the perception of recovery by the patient.
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia in the form of morphine 0.05 mg/kg will be given when the Visual Analogue Scale (VAS) is more than 3, with a total maximum of 20mg morphine / 24hrs.
Time to independent movement | 24 hours postoperatively
  Time to independent movement defined as time from performing the intervention to be able independently mobile e.g. using the bathroom, care for the baby).
Incidence of complications | 24 hours postoperatively
  Incidence of complications such as nausea, vomiting, itching, urine retention, sedation (opioid sedation score), (respiratory depression (respiratory rate less than 8 breath per minute) and lower limb weakness will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.